CLINICAL TRIAL: NCT06692894
Title: Defining Inflammatory Biomarkers of Cardiovascular Disease in Patients With Myelodysplastic Syndromes
Brief Title: Defining Inflammatory Markers of Cardiovascular Disease in Patients With Myelodysplastic Syndromes
Status: Recruiting | Type: Observational
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Diego Adrianzen Herrera, Medical Oncologist, Assistant Professor, University of Vermont
Other Study IDs: STUDY00003256/UVMCC2406
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Myelodysplastic Syndromes, Adult
Keywords: Myelodysplastic Syndromes; Hematology
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be processed to test DNA from serum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Myelodysplastic syndromes: All participants will be in one group. Participants will by adults with Myelodysplastic syndromes. Blood will be taken at regular appointments that are part of standard care.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Blood will be collected from one cohort to identify potential blood biomarkers.

SUMMARY:
Why Is This Research Study Being Conducted?

* The study wants to find out why people with a type of blood cancer called myelodysplastic syndromes (MDS) are more likely to have heart problems like heart disease and stroke.
* Researchers also want to see if certain proteins related to inflammation in the body can help predict these heart issues in MDS patients.
* By understanding this better, researchers hope to find new ways to detect and manage heart disease risks in people with MDS

DETAILED DESCRIPTION:
What Is Involved in The Study?

* This study will follow patients with MDS over 6 months.
* Participants will come to the hospital for the first visit. Participants will learn about the study, sign papers to join the study, and share some basic health information. Participants will also give a blood sample of 10 milliliters after not eating overnight.
* After the first visit, participants will come back to the hospital once a week for 3 weeks to give more blood samples after fasting overnight.
* The study team will call participants the day before each scheduled blood draw to remind you of your appointment.
* Then participants will return to the hospital for another visits once a month for the next 5 months. Participants will talk about any changes in their health and give a blood sample at each visit.
* Participants won't get any treatment as part of this study, but their participation will help researchers learn how inflammation affects the health of people with MDS
* Researchers will collect a small amount of blood (6-10 mL) per visit
* These blood collections are a normal part of medical care and won't require participants to come in more often than usual. The frequency of visits will be part of the routine care for myelodysplastic syndrome at the cancer center. Extra blood will be collected during standard of care blood draws in the clinic.
* Sessions will take about 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed diagnosis of MDS by bone marrow biopsy morphology, using the 2022 World Health Organization (WHO) classification for myeloid neoplasms
* Eastern Cooperative Oncology Group (ECOG) performance status ≤3
* Expected survival of at least 6 months
* Ability to provide consent

Exclusion Criteria:

* Cases meeting 2022 WHO criteria of MDS with excess blasts 2 as initial diagnosis
* Hematopoietic stem cell transplantation expected within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with MDS diagnosed and treated at UVMMC will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Biologic Variability of Markers of Inflammation in the Blood | over 6 months
  The within- and between-person biologic variability of an inflammation proteome over a period of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No